CLINICAL TRIAL: NCT02059031
Title: A Two Part, Single-center, Randomized, Open-label, Crossover Study to Assess The Relative Bioavailability of New Tablet Formulations of GSK1265744 in Healthy Adult Subjects
Brief Title: A Study to Assess The Relative Bioavailability of New Tablet Formulations of GSK1265744 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 117020
Record Dates: First submitted 2014-02-06; First posted 2014-02-11 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: integrase inhibitor; pharmacokinetics; HIV; relative bioavailability; food; GSK1265744
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A (Experimental): In Part A, subjects will be randomized to receive two new formulations of GSK1265744 30 mg (New formulation 1 -micronized [B], New formulation 2un-micronized [C]) and the sodium salt reference formulation 30 mg (Reference formulation [A]) in one of six sequences; ABC, BCA, CAB, BAC, ACB, CBA in three treatment periods under fasting condition.
  Interventions: Drug: GSK1265744 Reference formulation; Drug: GSK1265744 New formulation 1; Drug: GSK1265744 New formulation 2
- Part B (Experimental): Fifteen eligible subjects completing the Part A of the study will enter in to Part B where they will receive either formulation B or C. The selected drug (B or C) will be administered under fed (moderate fat meal) condition in the fourth treatment period.
  Interventions: Drug: GSK1265744 New formulation 1; Drug: GSK1265744 New formulation 2

INTERVENTIONS:
Drug: GSK1265744 Reference formulation — GSK1265744 (micronized) reference formulation is available as 30 mg tablet to be orally administered with 240 mL of water
  Arms: Part A
Drug: GSK1265744 New formulation 1 — GSK1265744 (micronized) New formulation 1 is available as 30 mg tablet to be orally administered with 240 mL of water
Drug: GSK1265744 New formulation 2 — GSK1265744 (un-micronized) New formulation 2 is available as 30 mg tablet to be orally administered with 240 mL of water

SUMMARY:
This study will evaluate two new GSK1265744 sodium salt tablet formulations and provide data for selection of one of these tablet formulations for use in Phase 3. This is a single-center, randomized, two part, open-label, crossover study in healthy adult subjects. Part A is a randomized, open-label, 3-way balanced cross-over design in 24 subjects to assess the oral bioavailability of two GSK1265744 sodium salt tablet formulations relative to the current GSK1265744 sodium salt formulation being used in the phase IIb studies under fasting conditions. Part A treatment periods will be separated by a 14 day washout. After completion of Part A, preliminary PK data will be analyzed and a decision will be made based on pre-specified criteria, as to which formulation will be used to conduct Part B. Fifteen subjects who will have participated in Part A will participate in Part B and receive the selected formulation with a moderate fat meal. All treatments will be administered as single 30 mg doses of GSK1265744. Safety evaluations and serial PK samples will be collected during each treatment period. A follow-up visit will occur 10 - 14 days after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Male and females aged between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* Body weight >= 50 kilogram (kg) and body mass index (BMI) within the range 18.5-31.0 kg/meter^2 (inclusive).
* A female subject is eligible to participate if she is of: non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy [for this definition, "documented" refers to the outcome of the investigator's/designee's review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records]; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 milli-international units per milliliter (MIU/mL) and estradiol < 40 picogram (pg)/ml (<147 picomole per liter [pmol/L]) is confirmatory]; child-bearing potential with negative pregnancy test as determined by a serum or urine human chorionic gonadotropin (hCG) test at screening or prior to dosing AND; agrees to use one of the contraception methods for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until the final study visit; OR has only same-sex partners, when this is her preferred and usual lifestyle.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in protocol. This criterion must be followed from the time of the first dose of study medication until 14 days post-last dose of study medication.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Alanine aminotransferase (ALT), alkaline phosphatase and bilirubin <= 1.5x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).

Exclusion Criteria:

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 grams of alcohol: 12 ounces (360 ml) of beer, 5 ounces (150 ml) of wine or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GlaxoSmithKline (GSK) Medical Monitor, contraindicates their participation.
* A history of regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency virus (HIV) antibody.
* The subject's systolic blood pressure is outside the range of 90-140 millimeter of mercury (mmHg), or diastolic blood pressure is outside the range of 45-90 mmHg.
* History of clinically significant cardiovascular disease including: exclusion criteria for screening ECG (a single repeat is allowed for eligibility determination) - Heart rate of <45 and >100 beats per minute for males and <50 and >100 beats per minute for females; QRS duration >120 milliseconds (msec); QT duration corrected for heart rate by Bazett's formula (QTc B) >450 milliseconds. Evidence of previous myocardial infarction (pathologic Q waves, S-T segment changes (except early repolarization); History/evidence of symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting (CABG) surgery or percutaneous transluminal coronary angioplasty (PCTA) or any clinically significant cardiac disease; Any conduction abnormality (including but not specific to left or right complete bundle branch block, AV block [2nd degree (type II) or higher], Wolf Parkinson White [WPW] syndrome); Sinus pauses > 3 seconds. Any significant arrhythmia which, in the opinion of the principal Investigator and GSK Medical Monitor, will interfere with the safety for the individual subject. Non-sustained (>=3 consecutive ventricular ectopic beats) or sustained ventricular tachycardia.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Part A: Composite of pharmacokinetic (PK) parameters to evaluate the relative bioavailability of GSK1265744 in the fasted state | Pre-dose, 0.5 hour(hr), 1hr, 2hrs, 3 hrs, 4 hrs, 6hrs, 8hrs, 12hrs, 24hrs (Day 2), 48hrs (Day 3), 72hrs (Day 4), 120hrs (Day 6) and 168hrs (Day 8) post dose
  PK parameters will include area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC[0-infinity]), AUC from time zero (pre-dose) to last time of quantifiable concentration within a subject across all treatments (AUC[0-t]), maximum observed concentration (Cmax) and concentration at 24h post-dose (C24)
Part B: Composite of PK parameters to evaluate the relative bioavailability of GSK1265744 in the fed state | Pre-dose, 0.5 hr, 1hr, 2hrs, 3 hrs, 4 hrs, 6hrs, 8hrs, 12hrs, 24hrs (Day 2), 48hrs (Day 3), 72hrs (Day 4), 120hrs (Day 6) and 168hrs (Day 8) post dose
  PK parameters will include AUC(0-infinity), AUC(0-t), Cmax and C24

SECONDARY OUTCOMES:
Part A: Composite of other PK parameters following administration of GSK1265744 in the fasted state | Pre-dose, 0.5hr, 1hr, 2hrs, 3 hrs, 4 hrs, 6hrs, 8hrs, 12hrs, 24hrs (Day 2), 48hrs (Day 3), 72hrs (Day 4), 120hrs (Day 6) and 168hrs (Day 8) post dose
  Other PK parameters will include apparent terminal phase half-life (t1/2), absorption lag time (tlag), time to Cmax (tmax), the percentage of AUC(0-infinity) obtained by extrapolation (%AUCex), time of last measurable concentration (tlast) and apparent oral clearance (CL/F)
Part A: Safety and tolerability parameters, including adverse events, concurrent medication, clinical laboratory screens, ECG, and vital signs assessments | Up to 13 weeks
  Clinical laboratory screens will include haematology, clinical chemistry and urinalysis. Vital sign assessment will include systolic and diastolic blood pressure and heart rate
Part B: Composite of other PK parameters following administration of GSK1265744 in the fed state | Pre-dose, 0.5 hr, 1hr, 2hrs, 3hrs, 4hrs, 6hrs, 8hrs, 12hrs, 24hrs (Day 2), 48hrs (Day 3), 72hrs (Day 4), 120hrs (Day 6) and 168hrs (Day 8) post dose
  Other PK parameters will include t1/2, tlag, tmax, %AUCex, tlast and CL/F
Part B: Safety and tolerability parameters will include adverse events, concurrent medication, clinical laboratory screens, ECG, and vital signs assessments | Up to 18 weeks
  Clinical laboratory screens will include haematology, clinical chemistry and urinalysis

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Overland Park, Kansas, United States